CLINICAL TRIAL: NCT05173935
Title: Complications Associated With Primary Placement of Radiologically-Inserted Gastrostomy Versus Percutaneous Endoscopic Gastrostomy for Feeding
Brief Title: Complications Associated With Primary Placement of Gastrostomy for Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Melissa J. Neisen, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 16-010077
Record Dates: First submitted 2021-11-29; First posted 2021-12-30 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Gastrostomy Tube
Keywords: complication; quality of life; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants are randomized to receive either RIG or PEG. Investigator and Outcomes Assessors are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG Group (Active Comparator): Subjects will gastrostomy tube placement via percutaneous endoscopic gastrostomy (PEG) method.
  Interventions: Procedure: Percutaneous endoscopic gastrostomy
- RIG Group (Active Comparator): Subjects will have the placement of a gastrostomy tube via radiologically-inserted gastrostomy (RIG) method.
  Interventions: Procedure: Radiologically-inserted gastrostomy

INTERVENTIONS:
Procedure: Percutaneous endoscopic gastrostomy — Gastrostomy tube placement using an endoscopic camera inserted via the mouth into the stomach to place the tube.
  Arms: PEG Group
Procedure: Radiologically-inserted gastrostomy — Gastrostomy tube placement using a temporary nasogastric tube placed from nose to stomach and fluoroscopy (x-rays).
  Arms: RIG Group

SUMMARY:
The purpose of the study is to compare pain, complications, and quality of life after gastrostomy tube is placed by either percutaneous endoscopic gastrostomy (PEG) or radiologically-inserted gastrostomy (RIG) method.

DETAILED DESCRIPTION:
Objectives:

Primary objectives: to assess 1) pain and 2) major and minor complications with gastrostomy-tube placement, comparing RIG with PEG

Secondary objectives:

* To compare costs associated with each technique
* To compare anesthesia type used with each technique
* To assess patient quality of life before and after the procedure

Co-primary outcome measures:

Efficacy Outcome - Trajectory of the average pain score (question 3, Cleeland Brief Pain Inventory) through Week 6

Statistical Null Hypothesis: The model-based estimates of the pain scores trajectories will be co-incident for the two placement approaches RIG compared to PEG.

Safety Outcome - Minor and major complication rate per participant

Statistical Null Hypothesis: The percentage of participants with at least one major or minor complication will be equal between RIG and PEG groups

Methods:

All participants meeting criteria for placement of gastrostomy tube for nutrition and not having any exclusion criteria will be prospectively randomized at the initial Home Enteral Nutrition (HEN) visit with physician, nurse and dietician. The randomization will be performed with the use of a 4-block randomization tool, based on the inclusion criteria and will not be intentionally matched for other demographics. Participants will be randomized to either undergo RIG with an Interventional Radiologist or PEG with a Gastroenterologist. Sixty-four participants will be randomized into each group for a total accrual of 128 patients. Participants will be randomized to receive one of two widely-accepted standards of care. The research component will involve the use of questionnaires during routine post-placement follow-up to assess for pain, quality of life, and complications.

Radiologic technique:

Radiologically-inserted gastrostomy (RIG) tubes are placed in one of three ways: either using 1) a balloon to dilate the tract without gastropexy T-fasteners, 2) a balloon to dilate the tract with gastropexy T-fasteners or 3) a peel-away sheath with gastropexy T-fasteners. All of the procedures occur in the interventional radiology procedural suite and are performed after informed consent is obtained. The participant receives weight-based antibiotics intravenously. A temporary small nasogastric or orogastric tube is placed if one is not in place. Suitable site for percutaneous access into the stomach is localized on the abdomen, sometimes with the use of ultrasound to mark the liver edge. Participants may or may not have had a CT scan of the abdomen for stomach localization prior to the placement. The abdomen is prepped and draped in the usual sterile fashion. Local anesthesia alone or with the addition of moderate sedation, monitored anesthesia care, or general anesthesia is administered, depending on the needs of the participant. Participant may or may not receive intravenous glucagon. Air is insufflated into the stomach through the nasogastric tube under fluoroscopic guidance. One percent lidocaine for local anesthesia is instilled at the desired gastrostomy site and at the sites of T-fasteners, if used. An 18-gauge or micropuncture needle is advanced into the insufflated stomach under fluoroscopic guidance. Air is aspirated, and contrast medium is injected to confirm the intraluminal location of the needle(s). A stiff guidewire is advanced into the stomach or through the stomach to the ligament of Treitz. For the balloon-dilatation technique, the tract is dilated with a balloon, the gastrostomy tube is advanced into the stomach using the balloon in coaxial fashion, and then the dilating balloon is removed. For the technique that uses a peel-away sheath, the tract is serially dilated over the wire, and a peel away sheath is advanced over the wire into the stomach. For both techniques, a 16- or 18-French balloon-style gastrostomy tube is then advanced into the stomach lumen, and the guide wire is removed. If T-fasteners are used, they are then secured to the participant's skin. T-fasteners are designed to fall off at six weeks. The nasogastric tube is removed at the end of the procedure. Participants may use the tube for water and medications at two hours and may use the tube for feedings no sooner than four hours, but only after appropriate Home Enteral Nutrition follow-up.

Endoscopic technique:

All PEG placements are performed with anesthesia support and after informed consent is obtained. After the participant is appropriately sedated and antibiotic prophylaxis is given, the standard adult gastroscope is passed orally and a routine esophagogastroduodenoscopy (EGD) is performed to assess for any unknown pathology and to characterize if appropriate apposition of the anterior gastric wall and the abdominal wall can be accomplished. This requires insufflation of air or carbon dioxide through the scope and then palpation of the abdominal wall and/or observation of the abdominal wall for light trans-illumination to identify the site of best apposition of the two walls. This site is marked and then cleansed. Local lidocaine is infiltrated and a small stab wound may be made at the discretion of the endoscopist. Using sterile technique a needle is passed through the abdominal wall into the gastric lumen as observed endoscopically. Through this needle is passed a looped flexible wire which is grasped with a snare introduced through the scope and the wire is withdrawn out the mouth as the scope is removed. A 20-French gastrostomy tube is attached to the looped wire and the wire is pulled from the abdominal wall so the tube is pulled through the mouth and down the esophagus into the stomach and out the abdominal wall. The tube is pulled into position until the inner bumper is noted to be at the abdominal wall. The faceplate is then placed over the external tube to maintain position. At the discretion of the endoscopist the scope may be passed once more into the stomach to ensure proper positioning of the tube. The tube may be used for fluid or feedings at 4 hours after initial placement, but only after appropriate Home Enteral Nutrition follow-up.

Independent of whether RIG or PEG is placed, the participants will be followed by the Home Enteral Nutrition clinic, using the following protocol:

1. Face-to-face visit with HEN nurse for site care and tube education and with HEN dietitian for instruction about provision of supplies and for administration of the first feeding together, to occur within 24 hours post-procedure.
2. Phone call or secure message at 48-86 hours post-procedure to answer questions and ensure proper progression of feeding.
3. Phone call or secure message or face-to-face visit 6 weeks post-procedure.
4. Face-to-face visit with HEN dietitian and nurse for tube exchange, at 3 months for RIG and 9 months for PEG, if needed, for first tube replacement.

Length of study: Participants will be followed until tube removed or until 9 months, whichever is shorter.

Data Collection:

Study data collected will include pain, major and minor complications, quality of life, rates of early exchange of tube, and costs associated with each procedure.

ELIGIBILITY:
Inclusion criteria:

* Age greater than or equal to 18 years
* Cannot maintain adequate nutrition by mouth

Exclusion criteria:

* Venting-only gastrostomy
* Patients with Amyotrophic Lateral Sclerosis (ALS)
* Coagulopathy with uncorrectable International Normalized Ratio (INR) greater than 1.5 or inability to hold anticoagulation
* Structural abnormality that would prevent one or both techniques

  * Known severe esophageal stricture
  * Obstructing malignancy in oropharynx or esophagus that prohibits pull-through technique
  * Neoplastic, inflammatory, or infiltrative disease of abdominal wall or gastric wall
  * Known hepatomegaly
  * Abdominal wall mesh
* Enteric functional abnormality

  * Small bowel or colonic obstruction
  * Gastric or small bowel dysmotility
* Active abdominal infection/peritonitis/enterocutaneous fistula
* Ascites
* Ventriculoperitoneal shunt
* Inpatient status
* Pregnant patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
Change in pain with gastrostomy-tube placement, comparing RIG with PEG | Before the procedure, within 24 hours after procedure, at 48-96 hours after procedure, and at 6 weeks after procedure
  Trajectory of the average pain score over time (question 3, Cleeland Brief Pain Inventory), which rates average pain in the past 24 hours, with 0 being no pain and 10 being pain as bad as can be imagined
Major and minor complications with gastrostomy-tube placement, comparing RIG with PEG | Within 24 hours after procedure
  Assessment of the following major complications after procedure: Peritonitis, Abscess, Major bleeding requiring intervention and/or transfusion, Bowel perforation, Death; Assessment of the following minor complications after procedure: Minor bleeding, not requiring transfusion, Tube occluded, Tube malpositioned/fell out,Tube damaged, Skin erosion, Site redness, Site nodules/induration, Site exudate
Major and minor complications with gastrostomy-tube placement, comparing RIG with PEG | At 6 weeks after procedure
  Assessment of the following major complications after procedure: Peritonitis, Abscess, Major bleeding requiring intervention and/or transfusion, Bowel perforation, Death; Assessment of the following minor complications after procedure: Minor bleeding, not requiring transfusion, Tube occluded, Tube malpositioned/fell out,Tube damaged, Skin erosion, Site redness, Site nodules/induration, Site exudate
Minor complications with gastrostomy-tube placement, comparing RIG with PEG | At 3 months, if tube still in place
  Assessment of the following complications after procedure: Tube occluded, Tube malpositioned/fell out, Tube damaged, Skin erosion, Site redness, Site nodules/induration, Site exudate
Minor complications with gastrostomy-tube placement, comparing RIG with PEG | At 6 months, if tube still in place
  Assessment of the following complications after procedure: Tube occluded, Tube malpositioned/fell out, Tube damaged, Skin erosion, Site redness, Site nodules/induration, Site exudate
Minor complications with gastrostomy-tube placement, comparing RIG with PEG | At 9 months, if tube still in place
  Assessment of the following complications after procedure: Tube occluded, Tube malpositioned/fell out, Tube damaged, Skin erosion, Site redness, Site nodules/induration, Site exudate

SECONDARY OUTCOMES:
Costs associated with gastrostomy tube placement, comparing RIG with PEG | Immediately after procedure completion
  Tally of costs associated.
Anesthesia type associated with gastrostomy tube placement, comparing RIG with PEG | Immediately after procedure completion
  Documentation of the types of anesthesia used during procedure
Patient quality of life associated with gastrostomy tube placement, comparing RIG with PEG, before and after the procedure | Before the procedure
  Measurement of the patient quality of life using the Short Form-8 Quality of Life (SF-8 QOL) inventory in which eight questions with five or six possible descriptive word answers exist, with the first answer of each question meaning a better outcome and the last answer of each question meaning a worse outcome
Patient quality of life associated with gastrostomy tube placement, comparing RIG with PEG, before and after the procedure | At 6 weeks after procedure
  Measurement of the patient quality of life using the Short Form-8 Quality of Life (SF-8 QOL) inventory in which eight questions with five or six possible descriptive word answers exist, with the first answer of each question meaning a better outcome and the last answer of each question meaning a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Neisen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials